CLINICAL TRIAL: NCT04664660
Title: Endometriosis and Risk Factors in Pregnancy, Labor and Delivery
Brief Title: Endometriosis and Obstetric Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Carlo Alboni, MD, PhD, Dr. Carlo Alboni MD, PhD Head of Minimally Invasive and Robotic Gynecologic Surgery Unit University Hospital of Modena - Italy, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: EndoPreg01
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Endometriosis; Obstetric Complication
Keywords: Endometriosis; Obstetric outcome; Delivery outcome; Neonatal outcome
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with previous histologic diagnosis of endometriosis
  Interventions: Other: Retrospective analysis of obstetrics outcomes
- Patient without endometriosis
  Interventions: Other: Retrospective analysis of obstetrics outcomes

INTERVENTIONS:
Other: Retrospective analysis of obstetrics outcomes — Retrospective analysis of clinical records including general medical and gynecological history, pregnancy course, delivery mode and newborn conditions.

SUMMARY:
The purpose of this study is to assess if endometriosis can be considered a risk factor for adverse obstetric and delivery outcomes

DETAILED DESCRIPTION:
This is a retrospective, observational, case-control study. Pregnancy, delivery and neonatal outcomes will be analyzed in two groups of patients (case and control group): women with diagnosis of endometriosis histologically confirmed and women without endometriosis. Women with endometriosis will be matched to controls by age. A database with general medical and gynecological history, pregnancy course, delivery mode and newborn conditions will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who delivered at Azienda Ospedaliero Universitaria Policlinico di Modena from 2000 to 2020
* Histologic diagnosis of endometriosis before pregnancy for case group
* Age matched healthy patients for control group

Exclusion Criteria:

* Clinical records not available

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who delivered at Azienda Ospedaliero Universitaria Policlinico di Modena from 2000 to 2020. Women with a histological diagnosis of endometriosis before pregnancy matched by age with healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Preterm delivery | Time of delivery
  Incidence of delivery before 37 weeks of pregnancy
Gestational diabetes | after 18 weeks' pregnancy
  fasting blood glucose >17 mmol/L
Gestational hypertension | after 20 weeks' gestation
  blood pressure persistently > 140/90 mm Hg
Assisted reproduction technologies | before pregnancy
  Patients who referred to assisted reproduction technologies
Cesarean Section | Time of delivery
  Robson Classifications
Postpartum hemorrhage | Time of delivery
  Greater than 500 mL estimated blood loss in a vaginal delivery or greater than 1000 mL estimated blood loss at the time of cesarean delivery
Birth-weight | Time of delivery
  small for gestational age (birth weight below the 10th percentile) or large for gestational age (birth weight over the 90th percentile)
Apgar scores | Time of delivery
  Apgar scores

CONTACTS AND LOCATIONS:
Locations (1):
- Carlo Alboni, Modena, Italy

IPD SHARING:
Plan to Share IPD: No
I prefer not to share individual participant data